CLINICAL TRIAL: NCT04350554
Title: Pregnancy in Women With HIV Infection: a Multicenter Cohort in Spain
Brief Title: Pregnancy in Women With HIV Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carlos III Health Institute (Other Government)
Collaborators: Red Temática de Investigación Cooperativa en Sida (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Inmaculada Jarrín Vera, Scientific, Carlos III Health Institute
Other Study IDs: RIS_EPICLIN_04_2020
Record Dates: First submitted 2020-04-09; First posted 2020-04-17 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections; Pregnancy Related
Keywords: HIV; Pregnancy; Adverse pregnancy outcomes
MeSH Terms: conditions — HIV Infections | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective pregnancies: Women recruited in CoRIS from January 2004 to November 2019 and who became pregnant during this period.
  Interventions: Other: Pregnancy
- Prospective pregnancies: Women recruited in CoRIS from January 2004 to November 2019 who will become pregnant during the year 2020 and who agree to participate in a telephone survey.
  Interventions: Other: Pregnancy

INTERVENTIONS:
Other: Pregnancy — To measure and characterize pregnancies and describe the clinical course during pregnancy
  Groups: Retrospective pregnancies
Other: Pregnancy — To evaluate attitudes towards pregnancy (ie. planned pregnancy) and social support among women who become pregnant during the year 2020
  Groups: Prospective pregnancies

SUMMARY:
Women living with HIV face multiple challenges regarding pregnancy, encompassing not only their intention to procreate, but also difficulties during the course of pregnancy.

Compared to HIV-negative controls, HIV-infected women have a higher risk of pregnancy complications such as preeclampsia, gestational diabetes, or preterm labor. In addition, the treatment of HIV among pregnant women entails specific difficulties, such as changes in bioavailability of antiretroviral drugs, or the concern about the association of certain antiretrovirals with adverse pregnancy outcomes.

There is very little evidence about pregnancy among women living with HIV in Spain. Very few studies have been published, performed in single centers or in small cohorts with a limited number of patients. The Cohort of the Spanish AIDS Research Network (CoRIS) offers a unique setting to answer questions that are unlikely to be answered by a single study.

The aims of this study are (i) to describe the incidence of pregnancies and their temporal trends from 2004 to 2019, (ii) o describe the clinical and epidemiological characteristics of women who become pregnant, (iii) to assess the diagnostic delay among women diagnosed with HIV infection after becoming pregnant, (iv) to investigate the clinical course during pregnancy and its predictive factors, (v) to describe the antiretroviral treatment administered to pregnant women, (vi) to describe clinical outcomes after pregnancy, (vii) to describe the outcome of the conception in terms of interrupted pregnancies, spontaneous abortions, term pregnancies, type of delivery (vaginal or caesarean section) and HIV infection of the newborn, and (vii) to evaluate attitudes towards pregnancy (ie. planned pregnancy) and social support among women who become pregnant during the year 2020.

Study population will be women from the cohort of the Spanish AIDS Research Network (CoRIS) who have become pregnant in the period 2004-2010.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive women recruited in CoRIS
* Became pregnant from January 2004 to November 2019
* or become pregnant during the year 2020 and agree to participate in a telephone survey

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The Cohort of the Spanish AIDS Research Network (CoRIS) is a prospective multicentre cohort of HIV-positive treatment-naïve patients aged >13 years, recruited from 46 centres from 13 Autonomous Regions in the Spanish public healthcare system. Recruitment and follow-up started in 2004 and are still ongoing. From 2004 to the last update in November 2018, 15,509 patients have been included in the cohort. This study will be performed using the update of November 2019, that will be available in June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of pregnancies | From 2004 to 2019
Epidemiological characteristics of women who become pregnant | 2004 to 2019
  Proportion of diagnostic delay among women diagnosed with HIV infection after becoming pregnant
Clinical course during pregnancy | 2004 to 2019
  Proportion of women with undetectable viral load at week 36 of pregnancy
Opportunistic infections during pregnancy | 2004 to 2019
  Incidence of opportunistic infections throughout pregnancy
Persistence of Antiretroviral treatment (ART) during pregnancy | 2004 to 2019
  Time from ART initition to treatment change during pregnancy
Antiretroviral treatment (ART) administered to pregnant women | 2004 to 2019
  Distribution of ART regimens administered to women at pregnancy
Follow-up after pregnancy | 2004 to 2019
  Rate of lost-to-follow-up during the first year after pregnancy termination
Clinical outcomes after pregnancy | 2004 to 2019
  Proportion of women with undetectable viral load 6 months after pregnancy termination
Outcome of the conception | 2004 to 2019
  Proportion of interrupted pregnancies, spontaneous abortions and term pregnancies
Term pregnancies | 2004 to 2019
  Proportion of term pregnancies
Type of delivery | 2004 to 2019
  Proportion of vaginal deliveries
HIV infection of the newborn | 2004 to 2019
  Proportion of newborns with HIV infections
Attitudes towards pregnancy | Pregnancies during the year 2020
  Proportion of unintended pregnancies (unplanned or unwanted at the time of conception)

IPD SHARING:
Plan to Share IPD: No
Data cannot be made publicly available because they are owned by a third party, the AIDs Research Network (RIS), and because participants agreed that data would only be used for research projects by RIS or those projects approved by its
  Executive and Scientific Committee. Interested readers may send requests for the data to proyectoscoris@gmail.com. Requests will be assessed by the Executive and Scientific Committee